CLINICAL TRIAL: NCT00437684
Title: A Pilot, Open Label, Multicenter, Randomized Clinical Trial on Lopinavir/Ritonavir-Monotherapy vs Lopinavir/Ritonavir Plus Selected Nucs, in HIV/HCV Coinfected Patients With Chronic Hepatitis C or Compensated Cirrhosis, Starting Treatment With Ribavirin and Pegylated Interferon
Brief Title: Lopinavir/Ritonavir Monotherapy Versus Standard Highly Active Antiretroviral Therapy (HAART) in HIV/HCV Coinfected Patients Starting Treatment With Anti-Hepatitis C Virus (HCV) Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Abbott (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Adriano Lazzarin, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kamon 2; NTC00437684
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections; Hepatitis C
Keywords: HIV/HCV; HIV and HCV coinfected patients; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Hepatitis C | interventions — Ribavirin

ARMS (2):
- A (Experimental): LPV/r: LPV/r monotherapy and anti HCV drugs for 12 months. All the patients will be followed-up for six months after the end of anti-HCV drugs for the evaluation of Sustained Virological Response (SVR). At the end of the co-treatment for HCV/HIV, each subject will be treated for HIV infection according to physician decisions.As anti-HCV drugs the patients will receive PEG-IFNa 2a 180 mcg/week + Ribavirin 1-1.2 g/day .At the end of the third month of combined therapy, only patients who reach an early virological response will continue anti-HCV drugs.
  Interventions: Drug: LPV/r; Drug: PEG-IFNa 2a; Drug: Ribavirin
- B (Active Comparator): LPV/r+ selected NUCS and anti HCV drugs for 12 months. All the patients will be followed-up for six months after the end of anti-HCV drugs for the evaluation of Sustained Virological Response (SVR). At the end of the co-treatment for HCV/HIV, each subject will be treated for HIV infection according to physician decisions.As anti-HCV drugs the patients will receive PEG-IFNa 2a 180 mcg/week + Ribavirin 1-1.2 g/day .At the end of the third month of combined therapy, only patients who reach an early virological response will continue anti-HCV drugs.
  Interventions: Drug: LPV/r; Drug: PEG-IFNa 2a; Drug: Ribavirin; Drug: NUCS

INTERVENTIONS:
Drug: LPV/r — 200/50 mg 2 cpr bid monotherapy
Drug: PEG-IFNa 2a — PEG-IFNa 2a 180 mcg/week
Drug: Ribavirin — Ribavirin 1-1.2 g/day
Drug: NUCS — Nucleoside Reverse Transcriptase Inhibitors
  Arms: B

SUMMARY:
The purpose of this study is to evaluate if the combination of Lpv/r monotherapy and anti-HCV drugs does not match with additional toxicity induced by the association of HAART and Peg-IFN + ritonavir in HIV/HCV coinfected patients.

Secondary objective is to assess if Lpv/r monotherapy during HCV-treatment is associated with HIV efficacy versus optimized HAART.

DETAILED DESCRIPTION:
This is a pilot, randomised, open label, controlled clinical trial. All eligible patients(CD4>350, HIV RNA<50 copies and no PI mutations) will be randomized (1:1) to receive LPV/r new tabs (200/50 mg, 2 cpr BID) monotherapy (arm A) or LPV/r + selected NUCS (arm B) associated to anti-HCV therapy for 12 months. The number of subjects to recruit, in each arm of the study, is equal to 25, the total number of subjects to enrol will be 50.

* Group A: will receive LPV/r monotherapy and anti HCV drugs for 12 months.
* Group B: will receive LPV/r+ selected NUCS and anti HCV drugs for 12 months. All the patients will be followed-up for six months after the end of anti-HCV drugs for the evaluation of Sustained Virological Response (SVR). At the end of the co-treatment for HCV/HIV, each subject will be treated for HIV infection according to physician decisions.As anti-HCV drugs the patients will receive PEG-IFNa 2a 180 mcg/week + Ribavirin 1-1.2 g/day .At the end of the third month of combined therapy, only patients who reach an early virological response will continue anti-HCV drugs.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >18 years old
* Subject has given written informed consent
* Subject has a confirmed diagnosis of HIV and HCV infection
* Subject is naive for HCV-infection treatment
* Subject has chronic hepatitis and/or subject has compensated cirrhosis (Child class A)
* Subject has a CD4+ count of > 350 cell/mmc
* Subject is HIV-RNA negative during the previous six month
* Subject is on stable HAART including r/LPV for > 6 months
* Subject has genotype available at baseline and no mutations associated with resistance to PI or no virologic failure on PI treatment, defined as a confirmed HIV-RNA level>50 cp/mL after 24 weeks, > 50 cp/ml after 48 weeks, or a repeated HIV RNA level > 50 cp/mL after prior suppression of viremia to< 50 cps/mL.
* Free of any clinically significant disease (other than HIV and HCV) that would interfere with study evaluations.
* Subject will use effective contraceptive methods for the duration of the study

Exclusion Criteria:

* Subject is HbsAg positive
* Subject has cirrhosis score Child-Pugh B/C,
* No previous hepatic decompensation
* Subject has HIV-related thrombocytopenia (Platelets count < 50.000/mmc)
* Subject has neutrophils count < 1500/mmc
* Subject has Hb value < 11 g/dL
* Subject has creatinine value > 1.5 mg/dL
* Subject is pregnant or wishes to become so
* Subject has any cause of liver disease other than chronic hepatitis C, status of liver decompensation or any other condition consistent with decompensated liver disease (bleeding from esophageal varices, signs of current bleeding, significant ascites, hepatic encephalopathy)
* Subject is alcohol abuser (> 30 gr/die)
* Subject has autoimmune hepatitis
* Prior treatment with PEG-IFN or ribavirin
* Illicit drugs abuse that in the opinion of the investigator could lead to poor compliance with the terms of the protocol (Methadone sostitution therapy allowed)
* Active heart disease (e.g. angina, congestive heart failure, recent myocardial infarction or significant arrhythmia)
* Subject has pre-existing severe depression, condition of severe psychiatric disorders such as suicidal ideation, suicide attempts, depression or acute psychosis
* Subject has uncompensated diabetes
* Subject has active opportunistic infections or major opportunistic infections during the previous 12 months
* Subject has known hypersensitivity or contraindication to study medications
* Subject has any other condition that in the opinion of the investigator will make the subject unsuitable for enrolment or will interfere with the subject participating in or completing the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-02; Primary Completion 2010-07 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To assess if the combination of LPV/r monotherapy in association with anti-HCV | 12 months
Nucs) and PEG-IFN alfa 2a +Ribavirin in patients naïve for HCV treatment | 12 months
without previous failure or detection of any mutations related to PI resistance. | 12 months

SECONDARY OUTCOMES:
To assess if LPV/r monotherapy during the HCV treatment is associated with | 12 and 18 months
anti HIV/HCV efficacy and a better patient satisfaction vs optimized HAART. | 12 and 18 months
To assess the number and type of HIV-1 resistance mutations in patients with | 12 and 18 months
virological failure | 12 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Lazzarin, MD, Principal Investigator — IRCCS San Raffaele Hospital
Locations (1):
- San Raffaele Hospital, Dep. Infectious Diseases, Milan, Italy

REFERENCES:
- [Derived] Hasson H, Galli L, Gallotta G, Neri V, Blanc P, D'Annunzio M, Morsica G, Sollima S, Merli M, Lazzarin A, Uberti-Foppa C. HAART simplification with lopinavir/ritonavir monotherapy in HIV/HCV co-infected patients starting anti-HCV treatment: a randomised pilot study (KaMon study). New Microbiol. 2012 Oct;35(4):469-74. Epub 2012 Oct 1. PMID 23109014